CLINICAL TRIAL: NCT05118217
Title: Retinal Microvascular Dysfunction in Non-Painful and Painful Diabetic Peripheral Neuropathy in Type 2 Diabetes Mellitus
Brief Title: Microvascular Dysfunction in Diabetic Peripheral Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Calvin Howorth, Principle Investigator/Lecturer of Podiatry, University of Plymouth
Other Study IDs: IRAS: 261329
Record Dates: First submitted 2020-10-12; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Peripheral Neuropathy; Painful Diabetic Neuropathy
Keywords: microvascular dysfunction; endothelial dysfunction
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical DPN without pain: * Score above 2.5 on the Michigan Neuropathy Screening Instrument
  * Score below 4 on the DN4
  Interventions: Other: This is a non-interventional study
- Painful DPN: * Score above 2.5 on the MNSI
  * Score above 4 on the DN4
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study

SUMMARY:
This study primarily seeks to evaluate dysfunction of small blood vessels and their linkage to dysfunction of nerves in people with Type 2 Diabetes. The purpose of this research is to explore some of the underlying pathophysiology of diabetic peripheral neuropathy, particularly painful diabetic peripheral neuropathy. The pain experienced by individuals with painful diabetic peripheral neuropathy is severe and associated with low quality of life. The pain does not typically respond well to pharmacological management. The processes underpinning the sources of pain are poorly understood, consequently only around a third of patients benefit from existing treatments. Some historic research on the sources of pain suggest the retention of the ability to reduce blood flow in small vessels may underpin these pain pathways. This research aims to explore this possibility, looking at the nerve-linked response in small vessels with a flickering light within the eye.

Participants will complete three or four questionnaires: one demographic, two to aid with stratifying participants into groups concerning symptoms of neuropathy and an additional questionnaire if participants are stratified to the painful DPN group. A basic neurological examination of the feet will follow.

Basic measurements of height, weight and blood pressure will be recorded for each participant.

The primary sites of measurement of this small vessel dysfunction will be the eye and the foot investigated in a non-invasive manner. A bright flickering light will be shone into participants eyes, with the reaction of small vessels recorded. Sensors will also be placed on the feet and chest of participants and warmed to ~44C. An image will be taken of participants eyes to measure nerve layer thickness and an area of skin on the forearm will be illuminated to measure for levels of a metabolic marker. A picture of the eye will also be taken to determine nerve layer thickness.

DETAILED DESCRIPTION:
This cross-sectional observational study will take place between November 2021 and May 2022 and will recruit individuals with Type 2 Diabetes alongside painful or non-painful peripheral neuropathy. The study aims to determine the relationship between microvascular and metabolic markers and i) clinical neuropathy, ii) of painful neuropathy and iii) severity of neuropathic pain within a Type 2 Diabetic cohort.

This will be done through achieving the following objectives:

i) determination of whether retinal vasodilation in response to flicker-light stimulus is associated with i) the severity of neuropathy, ii) the presence of painful neuropathy and iii) severity of neuropathic pain within a T2DM cohort.

ii) determination of whether levels of tissue-bound advanced glycation endproducts (AGEs) measured by skin autofluorescence are associated with i) the severity of neuropathy, ii) the presence of painful neuropathy and iii) severity of neuropathic pain within a T2DM cohort.

iii) determination of whether pedal skin transcutaneous oxygen tension (TcPO2) measured by transcutaneous oximetry is associated with i) the severity of neuropathy, ii) the presence of painful neuropathy and iii) severity of neuropathic pain within a T2DM cohort.

iv)determination of whether retinal nerve layer thickness is associated with the severity of neuropathy, the presence of painful neuropathy and severity of neuropathic pain within a T2DM cohort v)determination of whether the following factors are associated with the severity of neuropathy, the presence of painful neuropathy and severity of neuropathic pain within a T2DM cohort

* HbA1c
* Lipid profile
* Body Mass Index
* Blood Pressure

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above.
* Diagnosed with Type 2 Diabetes Mellitus (confirmed on clinical notes)
* History of an abnormal neurovascular testing result (typically, 10g monofilament test)
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.
* Must be willing to refrain from caffeine and tobacco consumption 24hrs before procedures are undertaken.
* Participants must be willing and able (in the Investigator's opinion) to undertake DN4, Brief Pain Inventory-DPN and Michigan Neuropathy Screening Instrument questionnaires.
* Able to lie flat

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Patients with neuropathy due to other aetiological causes, such as hereditary, metabolic, inflammatory, cervical and lumbar spine diseases; cerebrovascular diseases; uremia; alcohol use; or toxic factors.
* All patients with Type 1 diabetes.
* A positive history of malignancy; connective tissue or infectious disease;
* Deficiency of vitamin B12 or folate;
* Chronic renal failure;
* Liver failure;
* Glaucoma;
* Age-related macular degeneration
* Epilepsy;
* Severely sight-impaired
* Presence of a neurological disorder;
* Inflammatory arthropathies
* Pregnancy.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with Type 2 Diabetes and Diabetic Peripheral Neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2021-11-18 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic Vessel Analysis | during the procedure
  Retinal vasodilation in response to flicker light stimulus - Response will be recorded as baseline corrected flicker response (bFR). Baseline will be recorded as the period from -30 to -5 seconds prior to flicker light stimulation. bFR will be calculated as the difference between peak dilation after provocation (dil%) and the minimum of the subsequent reactive constriction (constr%) and the width of the baseline amplitude (width BL%).

SECONDARY OUTCOMES:
Static Vessel Analysis | during the procedure
  The standard parameters for Static Retinal Vessel Function observed will be as follows:
  * Diameter of the central retinal artery equivalent (CRAE)
  * Diameter of the central retinal vein equivalent (CRVE)
  * The ratio of CRAE-CRVE expressed as the arterio-venous ratio (AVR)
  Outcome Measure: AVR
Retinal Nerve Layer Thickness | during the procedure
  A measure of central retinal nerve fibre layer (RNFL) thickness will be obtained using the Heidelberg Spectralis OCT. This is a commercially available, non-invasive device that provides a high resolution scan of the retinal layers.
  Outcome Measure: Retinal Nerve Layer Thickness
Skin Autofluorescence | during the procedure
  Outcome Measure: Skin Autofluorescence (AU)
Transcutaneous Oximetry | during the procedure
  TcPO₂ (mmHg)
Blood pressure | during the procedure
  mmHg
Lipid Profile | pre-procedure
  HDL and LDL lipid levels - obtained from participants general practitioner with consent
HbA1c | pre-procedure
  As standard - obtained from participants general practitioner with consent
Body Mass Index | during the procedure
  Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Howorth, BSc (Hons), Principal Investigator — University of Plymouth

IPD SHARING:
Plan to Share IPD: Undecided
The Chief Investigator will have access to the final dataset. Any study data arising from the conduction of the study will be owned by the Sponsor (University of Plymouth). At the end of trial, anonymised participant level data may be shared with other researchers under an appropriate data sharing agreement. Data shared in this manner will ensure that the identity of all participants are obscured, and anonymity is enshrined in its presentation.